CLINICAL TRIAL: NCT01844323
Title: A Phase 1, Open-Label 4 Sequence 4 Period Crossover Study In Healthy Volunteers To Estimate The Effect Of Active Pharmaceutical Ingredient Particle Size And Lubrication On The Bioavailability Of A Single 125 Mg Dose Of Palbociclib (PD-0332991) Administered Under Fasted Conditions
Brief Title: A Study In Healthy Volunteers To Estimate The Effect Of The Active Ingredient Particle Size And Percentage Of The Excipients Used To Formulate The Capsules In The Dissolution Rate Of The Formulations In The Gastrointestinal Tract
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A5481022
Record Dates: First submitted 2013-04-16; First posted 2013-05-01 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Active Comparator): treatment A, reference, 20 micron palbociclib and lubrication level 1
  Interventions: Other: Palbociclib Formulation Reference
- Treatment B (Active Comparator): treatment B, test, 50 micron palbociclib and lubrication level 1
  Interventions: Other: Palbociclib Formulation Test
- Treatment C (Active Comparator): treatment C, test, 20 micron palbociclib and lubrication level 2
  Interventions: Other: Palbociclib Formulation Test
- Treatment D (Active Comparator): treatment D, test, 20 micron palbociclib and lubrication level 3
  Interventions: Other: Palbociclib Formulation Test

INTERVENTIONS:
Other: Palbociclib Formulation Reference — Single 45 mg dose; Dosage form is capsule taken orally.
  Arms: Treatment A
Other: Palbociclib Formulation Test — Single 45 mg dose; Dosage form is capsule taken orally.
  Arms: Treatment B
Other: Palbociclib Formulation Test — Single 45 mg dose; Dosage form is capsule taken orally.
  Arms: Treatment C
Other: Palbociclib Formulation Test — Single 45 mg dose; Dosage form is capsule taken orally.
  Arms: Treatment D

SUMMARY:
The particle size of the active ingredient may impact dissolution rate in the gastro intestinal tract and hence the amount of drug available for absorption. Similarly, differences in the percentage of the excipients used in the formulated capsules may affect dissolution rate. The purpose of this study is to estimate the effect that particle size and percentage of excipients could have in drug absorption, which will improve the manufacturing process of the formulated capsules.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or female subjects with no physical possibility of getting pregnant.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) preceding the first dose of study medication.
* Pregnant females; breastfeeding females; females with physical possibility of getting pregnant .

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Area under the Concentration-Time Curve (AUC) from time zero extrapolate to infinite time | 7 days
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 7 days
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Maximum Observed Plasma Concentration (Cmax) | 2 days

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 7 days
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area under the Concentration-Time Curve (AUC) from 0 to 72 | 3 days
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Apparent Oral Clearance (CL/F) | 7 days
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 2 days
Apparent Volume of Distribution (Vz/F) | 7 days
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Plasma Decay Half-Life (t1/2) | 7 days
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481022&StudyName=A%20study%20In%20Healthy%20Volunteers%20To%20Estimate%20The%20Effect%20Of%20The%20Active%20Ingredient%20Particle%20Size%20And%20Percentage%20Of%20The%20Excipients%20Used%20To